CLINICAL TRIAL: NCT05238961
Title: Neuroinflammation in Asymptomatic Carotid Artery Disease - Imaging Substudy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, Official Title: M.D. P.h.D., Director for the Division Molecular Imaging and Therapeutics Affiliation: University of Alabama at Birmingham, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R22-019
Record Dates: First submitted 2022-02-07; First posted 2022-02-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Critical Asymptomatic Carotid Artery Disease; Non-Critical Asymptomatic Carotid Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Critical Asymptomatic Carotid Stenosis Group (Experimental): Critical Stenosis Group: Diagnosis of Asymptomatic Carotid Artery Disease (aCAD) with >70% stenosis or peak systolic velocity on duplex ultrasound (DUS) ≥ 230 cm/s plus computed tomography angiography (CTA) or magnetic resonance angiography (MRA) confirmation.
  Interventions: Drug: [18F]DPA-714
- Cohort 2 - Controls-Non-Critical Asymptomatic Carotid Stenosis Group (Experimental): <40% carotid stenosis No planned revascularization
  Interventions: Drug: [18F]DPA-714

INTERVENTIONS:
Drug: [18F]DPA-714 — Investigational PET Tracer [18F]DPA-714

SUMMARY:
This clinical imaging substudy will use the small molecule translocator protein (TSPO) ligand, Fludeoxyglucose(18F)-labeled DPA-714, to compare neuroinflammation in individuals with high or low grade asymptomatic carotid artery stenosis (aCAD) who are participating in the separate Neuroinflammation in Asymptomatic Carotid Artery Disease study lead by Dr. Ron Lazar (IRB-300007806). The positron emission tomography (PET) tracer [18F]DPA-714 binds to the 18 kDa translocator protein (TSPO, also known as the peripheral benzodiazepine receptor) in the mitochondria of activated microglia/macrophages and provides a non-invasive measure of neuroinflammation.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 - Critical Asymptomatic Carotid Stenosis Group Inclusion Criteria:

1. Critical Stenosis Group: Diagnosis of Asymptomatic Carotid Artery Disease (aCAD) with >70% stenosis or peak systolic velocity on DUS ≥ 230 cm/s plus CTA or MRA confirmation.
2. Participation in University of Alabama at Birmingham (UAB) IRB protocol "Neuroinflammation in Asymptomatic Carotid Artery Disease" (IRB-300007806, PI Lazar).
3. Male or female age >18 years
4. English speaking with at least 8th grade education
5. High affinity binder for TSPO ligands based on genotyping for single nucleotide polymorphism (SNP) rs6971
6. Planned revascularization for aCAD in >14 days from time of consent

Cohort 2 - Non-Critical Asymptomatic Carotid Stenosis Group Inclusion Criteria:

1. Participation in UAB IRB protocol "Neuroinflammation in Asymptomatic Carotid Artery Disease" (IRB-300007806, PI Lazar).
2. <40% carotid stenosis
3. No planned revascularization
4. Male or female age 18 or older
5. English speaking with at least 8th grade education
6. High affinity binder for TSPO ligands based on genotyping SNP rs6971

Exclusion Criteria:

1. Contraindication to MRI
2. Pregnancy or lactation
3. Previous revascularization for treatment of aCAD
4. Prior stroke
5. Severe anemia (blood hemoglobin ≤ 8 mg/dL)
6. Previously obtained MRI scan with evidence of clinically significant abnormality
7. History of traumatic head injury defined by loss of consciousness >30 minutes or seizure at the time of the injury
8. Major depression
9. Known history of dementia
10. Serious medical comorbidity that, based on the judgement of the principal investigator, may interfere with study participation
11. Low or mixed-affinity binding for TSPO ligands based on genotyping for SNP rs6971.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2028-04-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Total volume distribution of the regional time-activity curves from the TSPO- PET Data. | Pre-study to 48 hours post PET imaging.
  The regional time-activity curves from the TSPO-PET data will be combined with image derived input function to provide estimates of total volume distribution (VT) based on a 2-tissue-compartment model (2-TCM) and graphical Logan plot analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD,PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States